CLINICAL TRIAL: NCT02876341
Title: Evaluating the Effect of Chronic Antihypertensive Therapy on New Onset Atrial Fibrillation and Clinical Outcomes in Septic Shock
Brief Title: Effects of Chronic Antihypertensive Therapy on Clinical Outcomes in Septic Shock
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16081002
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation; Septic Shock
Keywords: Chronic antihypertensives; New onset atrial fibrillation; Septic shock
MeSH Terms: conditions — Atrial Fibrillation; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No chronic antihypertensives: Not on either a chronic β-blocker or ACE-Inhibitor
- Chronic antihypertensives: On a chronic β-blocker, on chronic ACE-Inhibitor, or on both chronic β-blocker and ACE-inhibitor

SUMMARY:
Retrospective two-cohort study to determine the effect of chronic antihypertensive therapy on new onset atrial fibrillation and clinical outcomes in septic shock.

DETAILED DESCRIPTION:
This will be a retrospective two-cohort study to determine the effect of chronic antihypertensive therapy on new onset atrial fibrillation and clinical outcomes in septic shock. The two cohorts will be septic shock patients that were: 1) not on either a chronic β-blocker or angiotensin-converting-enzyme inhibitor (ACE inhibitor) or 2) on a chronic β-blocker, on chronic ACE-Inhibitor, or on both chronic β-blocker and ACE-inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older
* Diagnosis of septic shock requiring vasopressor therapy (norepinephrine, epinephrine, phenylephrine, dopamine, or vasopressin)
* Admitted to the medical intensive care unit (MICU) at Rush University Medical Center (RUMC)
* Time frame: 01/01/2012 to 07/1/2016

Exclusion Criteria:

* Pregnant patients
* Transfer from outside hospital on vasopressors
* Admitted to MICU in cardiopulmonary arrest
* Prior arrest within 24 hours of admission to RUMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, non pregnant medical intensive care (MICU) patient's with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Cumulative percent (%) of patients with new onset atrial fibrillation at 48 hours | 48 hours
  New onset atrial fibrillation defined as atrial fibrillation not present on admission to MICU

SECONDARY OUTCOMES:
Heart rate > 100 | 48 hours
  Total number of times with heart rate greater than 100 in 48 hours.
New onset of other arrhythmias | 48 hours
  Total onset of other arrhythmias not present on admission. Examples include, ventricular fibrillation, ventricular tachycardia, heart blocks, etc
Peak lactate | 48 hours
  Peak lactate level during the first 48 hours of admission
Duration of mechanical ventilation | During admission
In hospital mortality | During admission
28 day mortality | 28 days after discharge
90 day mortality | 90 days after discharge
New onset atrial fibrillation for patients on other antiarrhythmics | 24 and 48 hours
  Antiarrhythmic agents that are used to suppress abnormal rhythms of the heart (cardiac arrhythmias), such as atrial fibrillation, atrial flutter, ventricular tachycardia, and ventricular fibrillation. Will include any single or combination of class I, II, III, IV antiarrhythmic agents
Cumulative percent (%) of patients with new onset atrial fibrillation at 24 hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joshua DeMott, Pharm.D., Principal Investigator — Rush University Medical Center; Ishaq Lat, Pharm.D., Principal Investigator — Rush University Medical Center; Gourang Patel, Pharm.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush Univeristy Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined